CLINICAL TRIAL: NCT06116123
Title: Comparison of the Pressure Ulcer Prevention Effects of Two Mattresses With Different Support Surfaces Used in Bedridden Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Agri Ibrahim Cecen University (Other)
Responsible Party: Principal Investigator, Ramazan DENİZ, Principal Investigator, Agri Ibrahim Cecen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ataturk university
Record Dates: First submitted 2023-10-25; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Pressure Ulcer; Nursing Caries
MeSH Terms: conditions — Pressure Ulcer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Massage mattress with cube/block system) (Experimental)
  Interventions: Device: Massage mattress with cube/block system
- Group II (Standard of care) (No Intervention)

INTERVENTIONS:
Device: Massage mattress with cube/block system — Patients with an odd number were assigned to group I, while those with an even number were allocated to group II. Patients in group I were provided with a pressure sore prevention bed featuring a support surface with vibration (massage) capabilities, a cube/block system creating a low-pressure area, and a ventilation system, routinely utilized in the unit. For group II patients, a viscoelastic pressure sore prevention mattress with an orthopedic support surface, routinely employed in the unit, was used.Within the first six hours after admission, patients in both groups underwent initial assessments using the Braden Scale to determine their pressure sore risk. Both groups were monitored for a maximum of four weeks, with daily pressure ulcer assessments conducted using the Pressure Ulcer Observation Form. Pressure sore area in both groups was calculated in square centimeters (cm2) using the Wound Measurement Ruler.
  Arms: Group I (Massage mattress with cube/block system)

SUMMARY:
Aim: This study was conducted to investigate the effectiveness of two types of mattresses with different support surfaces used in bedridden patients.

Method: The sample of this quasi-experimental study consisted of 60 patients according to the inclusion criteria. A group I and group II of 30 patients each were formed from the sampled patients. For the patients in group I, a bed with a cube/block system and vibration (massage) feature was used. For the patients in group II, a viscoelastic mattress was used. The data of the study were collected with the ''Patient Identification Form'', ''Braden Scale'', ''Pressure Wound Observation Form'' and ''Wound Measurement Chart''. Number-percentage distributions, Chi-square, Fisher's Exact Probability Test and Mann-Whitney-U tests were used to evaluate the data.

Implications for Clinical Practice: It was determined that the support surface used affected the pressure sore size and the mattress with cube/block system and vibration (massage) feature created smaller sized wounds in the sacrum, trochanter, malleolus and heel regions. In the sacrum, scapula, and heel regions, although not statistically significant in terms of wound stage and the number of patients who developed pressure sores, it was seen that the mattress with cube/block system and vibration (massage) feature was more effective.

ELIGIBILITY:
Inclusion Criteria:

* A "low risk" rating on the Braden Scale.
* Voluntary informed consent from conscious patients and consent from the legal guardian for unconscious or confused patients.
* Absence of pressure sores upon admission to the clinics.
* A BMI (Body Mass Index) not exceeding 30.00 (as classified by the World Health Organization).

Exclusion Criteria:

* The patient's bed was changed in less than ten days after inclusion in the study,
* Patient referral,
* Discharge
* Exhitus was the exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2021-09-12 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Number of patients without pressure ulcers | Patients were followed up for four weeks.
  The formation of pressure sores in patients will be prevented with a bed with cube/block system massage feature. The massage feature of the bed will be used for this. In addition, the pressure in the relevant area will be reduced by removing the cubes inside the bed.

CONTACTS AND LOCATIONS:
Locations (1):
- Agri İbrahim Cecen University, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No